CLINICAL TRIAL: NCT01261429
Title: Phase II Study of Nilotinib Efficacy in Pigmented Villo-Nodular Synovitis/ Tenosynovial Giant Cell Tumour (PVNS/TGCT)
Brief Title: Study of Nilotinib Efficacy in Pigmented Villo-Nodular Synovitis/ Tenosynovial Giant Cell Tumour (PVNS/TGCT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: David Pérol, Centre Léon Bérard, 28 rue Laënnec, 69373, Lyon
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PVNS; 2010-018869-29 (EudraCT Number)
Record Dates: First submitted 2010-12-15; First posted 2010-12-16 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Pigmented Villonodular Synovitis
Keywords: Pigmented villonodular synovitis; tenosynovial giant cell tumour; nilotinib
MeSH Terms: conditions — Synovitis, Pigmented Villonodular | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nilotinib (Experimental)
  Interventions: Drug: Tasigna

INTERVENTIONS:
Drug: Tasigna — The study drug is nilotinib (Tasigna®). All patients will be administered with nilotinib 400 mg twice a day for one year. The patient will begin the treatment the day of inclusion.
  The prescribed dose should be swallowed whole with a glass of water. Doses of 400 mg should be administered twice daily approximately 12 hours apart. Patients should not eat within two hours before and one hour after taking nilotinib and need to avoid foods such as grapefruit juice which may inhibit CYP3A4 enzymes.

SUMMARY:
The purpose of this study is to explore the efficacy of nilotinib as a treatment of patients with progressive or relapsing pigmented villo-nodular synovitis / tenosynovial giant cell tumour (PVNS/TGCT) who cannot be treated by surgery.

The primary objective of the study will be to determine the efficacy of 12 weeks (3 months) of nilotinib treatment as measured by the non progression rate (Complete response + Partial Response + Stable disease according to Response Evaluation Criteria In Solid Tumours - RECIST version 1.1) in patients with progressive or relapsing PVNS/TGCT who cannot be treated by surgery.

this study is an international, multicentre, non-randomized, open-label phase II clinical trial with a Bayesian design.

A maximum sample size of 50 patients will be included in the study

DETAILED DESCRIPTION:
A key secondary objective of the study will be to determine the efficacy of 24 weeks (6 months) of nilotinib treatment as measured by the non progression rate (Complete response + Partial Response + Stable disease according to Response Evaluation Criteria In Solid Tumours - RECIST version 1.1) in patients with progressive or relapsing PVNS/TGCT who cannot be treated by surgery.

This key secondary objective was defined for the purpose of a further analysis (not described in this protocol) which will pool the data of the PVNS study with those of a similar concomitant study conducted in the US and Australia.

The other secondary objectives will be:

To evaluate the efficacy of nilotinib according to:

* The objective tumour response rate (Complete response + Partial Response according to RECIST version 1.1) after 12 weeks of treatment
* The duration of treatment response
* The best overall response obtained during the study
* The progression-free survival (PFS)
* The time to progression (TTP)
* The time to treatment failure (TTF)
* The proportion of patients with an operable tumour after nilotinib exposure according to investigator evaluation
* The description of concomitant treatments use
* The correlation between trough levels of nilotinib and objective tumour response To assess the safety of nilotinib for PVNS/TGCT patients

An exploratory objective of the study will be to study the relationship between the objective tumour response and the following tumour characteristics (tissues collected in a prior surgery, or by biopsy, upon specific acceptance by the patient; if no tissue is available in the prior surgery, a biopsy will be done at visit 2):

Presence of COL6A3/CSF1 fusion gene Presence of M-CSF, CSF1R, KIT, PDGFRA and B on immunohistochemistry Presence of phosphorylated c-fms on tumour samples Activation of the PI3K/Akt/mTor pathway, presence of activating mutations of ras, and other potential molecular alterations

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Histologically confirmed diagnosis of inoperable progressive or relapsing PVNS/TGCT OR resectable tumour requesting mutilating surgery
* Demonstrated progressive disease in the last 12 months
* At least one measurable site of disease on MRI/CT scan according to RECIST criteria (RECIST version 1.1) based on investigator's assessment
* WHO Performance status of 0, 1 or 2
* Adequate organ, electrolyte and marrow function, defined as the following: serum bilirubin > or =1.5 x ULN, ALT and AST < or = 2.5 x ULN, serum creatinine < or = 1.5 x ULN or creatinine clearance > or = 50 mL/min, absolute neutrophil count (ANC) > or = 1.5x109/L, platelets > or = 100x109/L, serum lipase < or =1.5 x ULN, magnesium ≥ lower limit of normal (LLN) and potassium ≥ LLN
* Prior adequate physical examination including weight, height, ECOG PS and vital signs (systolic and diastolic blood pressure, heart rate after at least 5 minutes in supine position)
* Signed written informed consent form
* Covered by a medical insurance (in countries where applicable)

Exclusion Criteria:

* Pregnant or lactating female or female of child-bearing potential not employing adequate contraception during the study and for up to three months following termination of the study
* Known hypersensitivity to nilotinib or to any of the excipients, galactose intolerance, lactase deficiency or glucose-galactose malabsorption prior to enrollment
* Acute or chronic uncontrolled liver disease, or severe renal disease
* Impaired cardiac function, including:
* LVEF<50% or below the institutional lower limit of the normal range (whichever is higher) as determined by echocardiogram or MUGA scan
* History or signs of prior myocardial infarction
* History of unstable angina
* Congenital long QT prolongation
* Personal history of unexplained syncope
* QTc interval ≥ 450 msec on screening ECG
* Other clinically significant heart disease (e.g. bradycardia, congestive heart failure or uncontrolled hypertension)
* Patient with family history of long QT syndrome, of unexplained syncope or of unexplained sudden death
* Patients with severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol e.g. uncontrolled diabetes, active or uncontrolled infection, history of pancreatitis
* History of non-compliance to medical regimens
* Concomitant treatment with medicinal products that induce CYP3A4 (e.g. dexamethasone, phenytoin, carbamazepine, rifampicin, phenobarbital or St. John's Wort), or that inhibit the CYP3A4 activity (e.g. ketoconazole, itraconazole, voriconazole, erythromycin, clarithromycin, telithromycin)
* Concomitant treatment with warfarin
* Concomitant treatment with anti-arrhythmic drug (e. g. amiodarone, sotalol, disopyramide, quinidine, procainamide) or medication that prolongs the QT interval (e.g. chloroquine, chlorpromazine, domperidone, droperidol, halofantrine, haloperidol, methadone, pentamidine, pimozide, thioridazine)
* Prior treatment with imatinib except if no progression was demonstrated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
the non progression rate after 12 weeks (3 months) of treatment, based on the response evaluated by CT scan or MRI according to RECIST criteria (RECIST version 1.1) and validated by a central review committee. | after 12 weeks (3 months) of treatment

SECONDARY OUTCOMES:
Non progression rate after 24 weeks (6 months) of treatment, based on the response evaluated by CT scan or MRI according to RECIST criteria (RECIST version 1.1). | after 24 weeks (6 months) of treatment
Objective tumour response according to RECIST version 1.1 (CR and PR) after 12 weeks of treatment | after 12 weeks of treatment
Duration of response | during the study
Best overall response | during the study
Progression-free survival | during the study
Time to progression | during the study
Time to treatment failure | during the study
Non progression rate after 12 weeks of treatment, based on the response evaluated locally by the investigator in charge using CT scan or MRI and according to RECIST criteria (RECIST version 1.1) | after 12 weeks of treatment
Proportion of patients with an operable tumour after nilotinib exposure according to investigator evaluation | at the end of the study (last visit)
Concomitant treatment use during the study | during the study
Correlation between trough level of nilotinib at 6 weeks and 12 weeks and objective tumour response | at the end of the study
Safety evaluation will be based on overall safety profile characterized by type, frequency and severity (as graded using NCI-CTCAE V3.0) of adverse events. | at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Jean Yves Blay, PR, Principal Investigator — Centre Léon Bérard, Lyon
Locations (15):
- France (8):
  - Institut Bergonié, Bordeaux
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital La Timone, Marseille
  - Institut Paoli Calmettes, Marseille
  - Institut Curie, Paris
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif
- Italy (2):
  - Istituto Nazionale dei Tumori, Milan
  - Regina Elena National Cancer Institute, Roma
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Radboud University Nijmegen Medical Centre, Nijmegen
- Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw, Poland
- United Kingdom (2):
  - University College Hospital UCL Hospitals NHS Foundation Trust, London
  - Oxford Cancer Centre, Oxford

REFERENCES:
- [Background] Mendenhall WM, Mendenhall CM, Reith JD, Scarborough MT, Gibbs CP, Mendenhall NP. Pigmented villonodular synovitis. Am J Clin Oncol. 2006 Dec;29(6):548-50. doi: 10.1097/01.coc.0000239142.48188.f6. PMID 17148989
- [Background] Martin RC 2nd, Osborne DL, Edwards MJ, Wrightson W, McMasters KM. Giant cell tumor of tendon sheath, tenosynovial giant cell tumor, and pigmented villonodular synovitis: defining the presentation, surgical therapy and recurrence. Oncol Rep. 2000 Mar-Apr;7(2):413-9. PMID 10671695
- [Background] West RB, Rubin BP, Miller MA, Subramanian S, Kaygusuz G, Montgomery K, Zhu S, Marinelli RJ, De Luca A, Downs-Kelly E, Goldblum JR, Corless CL, Brown PO, Gilks CB, Nielsen TO, Huntsman D, van de Rijn M. A landscape effect in tenosynovial giant-cell tumor from activation of CSF1 expression by a translocation in a minority of tumor cells. Proc Natl Acad Sci U S A. 2006 Jan 17;103(3):690-5. doi: 10.1073/pnas.0507321103. Epub 2006 Jan 6. PMID 16407111
- [Background] Cupp JS, Miller MA, Montgomery KD, Nielsen TO, O'Connell JX, Huntsman D, van de Rijn M, Gilks CB, West RB. Translocation and expression of CSF1 in pigmented villonodular synovitis, tenosynovial giant cell tumor, rheumatoid arthritis and other reactive synovitides. Am J Surg Pathol. 2007 Jun;31(6):970-6. doi: 10.1097/PAS.0b013e31802b86f8. PMID 17527089
- [Background] Dewar AL, Cambareri AC, Zannettino AC, Miller BL, Doherty KV, Hughes TP, Lyons AB. Macrophage colony-stimulating factor receptor c-fms is a novel target of imatinib. Blood. 2005 Apr 15;105(8):3127-32. doi: 10.1182/blood-2004-10-3967. Epub 2005 Jan 6. PMID 15637141
- [Background] Blay JY, El Sayadi H, Thiesse P, Garret J, Ray-Coquard I. Complete response to imatinib in relapsing pigmented villonodular synovitis/tenosynovial giant cell tumor (PVNS/TGCT). Ann Oncol. 2008 Apr;19(4):821-2. doi: 10.1093/annonc/mdn033. Epub 2008 Feb 21. No abstract available. PMID 18296418
- [Background] Brownlow N, Russell AE, Saravanapavan H, Wiesmann M, Murray JM, Manley PW, Dibb NJ. Comparison of nilotinib and imatinib inhibition of FMS receptor signaling, macrophage production and osteoclastogenesis. Leukemia. 2008 Mar;22(3):649-52. doi: 10.1038/sj.leu.2404944. Epub 2007 Sep 13. No abstract available. PMID 17851554
- [Background] P. A. Cassier, S. Stacchiotti, H. Gelderblom, D. M. Thomas, W. Van Der Graaf, B. M. Seddon, D. Julien, A. J. Wagner, J. Blay. Imatinib mesylate for the treatment of locally advanced and/or metastatic pigmented villonodular synovitis/tenosynovial giant cell tumor (PVNS/TGCT). J Clin Oncol. 2010 (suppl; abstr 10012); 28:15s. Meeting: 2010 ASCO Annual Meeting Abstract No: 10012
- [Background] V. Ravi, W. Wang, D. M. Araujo, J. A. Ludwig, R. J. Luke, V. O. Lewis, J. C. Trent, R. S. Benjamin, S. Patel. Imatinib in the treatment of tenosynovial giant-cell tumor and pigmented villonodular synovitis. J Clin Oncol. 2010 (suppl; abstr 10011); 28:15s. Meeting: 2010 ASCO Annual Meeting Abstract No: 10011
- [Derived] Spierenburg G, Grimison P, Chevreau C, Stacchiotti S, Piperno-Neumann S, Le Cesne A, Ferraresi V, Italiano A, Duffaud F, Penel N, Metzger S, Chabaud S, van der Heijden L, Perol D, van de Sande MAJ, Blay JY, Gelderblom H. Long-term follow-up of nilotinib in patients with advanced tenosynovial giant cell tumours: Long-term follow-up of nilotinib in TGCT. Eur J Cancer. 2022 Sep;173:219-228. doi: 10.1016/j.ejca.2022.06.028. Epub 2022 Aug 3. PMID 35932628
- [Derived] Gelderblom H, Cropet C, Chevreau C, Boyle R, Tattersall M, Stacchiotti S, Italiano A, Piperno-Neumann S, Le Cesne A, Ferraresi V, Penel N, Duffaud F, Cassier P, Toulmonde M, Casali P, Taieb S, Guillemaut S, Metzger S, Perol D, Blay JY. Nilotinib in locally advanced pigmented villonodular synovitis: a multicentre, open-label, single-arm, phase 2 trial. Lancet Oncol. 2018 May;19(5):639-648. doi: 10.1016/S1470-2045(18)30143-8. Epub 2018 Mar 20. PMID 29571946